CLINICAL TRIAL: NCT06726525
Title: Hydroxypropyl-methylcellulose and GlicoPro® Eyedrops in the Treatment of Dry Eye Disease: Clinical Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: FB VISION, Ascoli Piceno, Italy (Unknown); University of Messina (Other)
Responsible Party: Principal Investigator, Edoardo Villani, Associate professor of ophthalmology, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prot. 20-22
Record Dates: First submitted 2024-12-01; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye
Keywords: dry eye disease; GlicoPro®; Hydroxypropyl-methylcellulose
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HPMC+GlicoPro Group (Experimental)
  Interventions: Device: HPMC+GlicoPro eyedrops
- HPMC alone Group (Active Comparator)
  Interventions: Device: Hydroxypropyl-methylcellulose

INTERVENTIONS:
Device: HPMC+GlicoPro eyedrops — HPMC+GlicoPro eyedrops, artificial tears for dry eye disease
  Arms: HPMC+GlicoPro Group
Device: Hydroxypropyl-methylcellulose — Hydroxypropyl-methylcellulose eyedrops, artificial tears for dry eye disease
  Arms: HPMC alone Group

SUMMARY:
The goal of this clinical trial is to learn if Hydroxypropyl-methylcellulose and GlicoPro® eyedrops work to treat mild-to-moderate dry eye disease in adult patients. The main questions it aims to answer are:

Do Hydroxypropyl-methylcellulose and GlicoPro® eyedrops reduce patients' symptoms? Do Hydroxypropyl-methylcellulose and GlicoPro® eyedrops increase patients' tear film stability? Researchers will compare Hydroxypropyl-methylcellulose and GlicoPro® eyedrops to Hydroxypropyl-methylcellulose without GlicoPro® eyedrops to see if Hydroxypropyl-methylcellulose and GlicoPro® formulation works better to treat dry eye..

Participants will

* Take Hydroxypropyl-methylcellulose and GlicoPro® eyedrops or Hydroxypropyl-methylcellulose eyedrops every day for 3 months
* Visit the clinic 3 times in 3 months for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ocular Surface Disease Index (OSDI) >12 AND <65
* Fluorescein breakup time (FBUT) <10 seconds OR (Oxford staining Score >1 AND <4).

Exclusion Criteria:

* Systemic or ocular diseases with known effect on tear film and ocular surface
* Systemic or ocular medications with known effect on tear film and ocular surface
* Contact lens wearing,
* Ocular surgery in the 12 months before enrollment
* Known allergy or poor tolerance to any ingredient of the study products
* Presumed poor compliance to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) overall treatment effect | From enrollment to the end of treatment at 3 months
  OSDI is a standardized questionnaire for dry eye symptoms (Schiffman RM, et al. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. ).
  OSDI overall treatment effect (Month 1 and Month 3)
Symptom Assessment iN Dry Eye (SANDE) overall treatment effect | From enrollment to the end of treatment at 3 months
  SANDE is a validated short global dry eye symptom index (Schaumberg DA, et al. Development and validation of a short global dry eye symptom index. Ocul Surf. 2007 Jan;5(1):50-7) SANDE overall treatment effect (Month 1 and Month 3)
Fluorescein Break-up time (FBUT) overall treatment effect | From enrollment to the end of treatment at 3 months
  FBUT is a widely used method to assess tear film stability (Wolffsohn JS, et al. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. ) FBUT overall treatment effect (Month 1 and Month 3).

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Villani, MD, Study Director — University of Milan
Locations (1):
- Ophthalmology Clinic, Dept. of Biomedical Sciences, University of Messina, Messina, Italy, Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Villani E, Campagna G, Gentili V, Postorino EI, Genovese P, Palino P, Maini G, Carbucicchio A, Ferioli E, Nucci P, Rizzo R, Aragona P. Hydroxypropyl-Methylcellulose and GlicoPro(R) Eyedrops in the Treatment of Dry Eye Disease: In Vitro and Clinical Study. Ophthalmol Ther. 2025 Apr;14(4):787-803. doi: 10.1007/s40123-025-01101-6. Epub 2025 Mar 1. PMID 40024993